CLINICAL TRIAL: NCT03310996
Title: Use of Non-invasive Brain Stimulation for Working Memory Deficits in Neurofibromatosis Type 1
Brief Title: Non-invasive Stimulation in Neurofibromatosis Type 1
Acronym: tDCS is NF1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Shruti Garg, Dr, University of Manchester
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: SGIRAS21773
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Neurofibromatosis 1
Keywords: working memory
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: NeuroConn DC-STIMULATOR PLUS (NeurConn, GmbH), model number: 0021; serial number: 0351
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both sham and active treatment arms will have electrodes places on the scalp. The sham arm will have the current turned off in 10 seconds.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS Active arm (Experimental): The experimental arm will have the tDCS stimulation electrodes placed on the scalp and the current will be delivered over 20 minutes
  Interventions: Other: Transcranial direct current stimulation
- tDCS Sham arm (Placebo Comparator): The sham arm will have electrodes placed over the scalp and will be given the current for 10 seconds after which it will be ramped down and stopped.
  Interventions: Other: Transcranial direct current stimulation

INTERVENTIONS:
Other: Transcranial direct current stimulation — tDCS is an established research tool for non-invasive modulation of neuroplasticity. It has shown promise as a neurorehabilitation tool and demonstrated positive effects in various clinical conditions such as Alzheimer's, stroke, childhood psychosis, epilepsy and dystonias. tDCS uses low-intensity DC currents to modulate spontaneous neuronal network activity by altering the resting membrane potential.
  Other Names: Non-invasive brain stimulation

SUMMARY:
Intellectual impairments are a significant cause of morbidity in children with birth defects along with long term implication on academic and occupational functioning. Long lasting functional changes in the brain occur when children learn new things or memorise new information. Enhancing this and learning is a key objective inneurodevelopment and neuro-rehabilitation. This is pilot study aimed at testing a experimental neuroscience technique, Transcranial Direct Current Stimulation (tCDS) on the cognitive functioning of the brain in children with Neurofibromatosis type 1 (NF1). tDCS is an established research tool and has the potential for ameliorating the cognitive impairments associated with NF1. There is a growing interest in the use of tDCS in children but to our knowledge there have been no reported studies using tDCS intervention in NF1. 16 children aged 11-16 years will be recruited through the Manchester Centre of Genomic Medicine NF1 database. Participants will be randomised to receive active or sham tDCS. The treatment will be delivered for 20 minutes for 3 days. In the experimental group a 1mA current will be applied for 20 mins ; in sham tDCS the electrodes will be placed in an identical spot but the current is ramped down to 30 seconds to prevent stimulation. The aim of the study is to look into the acceptability and feasibility of using tDCS intervention within the NF1 group, obtain pilot data on the effect of tDCS on EEG (Electroencephalogram), cognitive and behavioural measures.

DETAILED DESCRIPTION:
16 children between the age of 11-16 years will be recruited through Manchester Centre of Genomic Medicine NF1 Database. The participants will be randomly assigned to 2 groups- active and sham treatment based on a computer generated random allocation list. The assessors will remain blind to treatment allocation.

On day 1, parents will be requested to complete well validated and standardised questionnaires. Baseline recording of the brain activity EEG(Electroencephalogram) will be measured and the baseline cognitive assessments will be completed on the participants. tCDS will be administered for 20 minutes alongside a simultaneous training task for working memory. Days 2, the tDCS (active or sham) will be delivered simultaneous with the training task for 20 minutes. On day 3, the tDCS intervention will be delivered followed by repeating the outcome measures similar to day 1.

A questionnaire investigating side-effects be will be completed by participant after each stimulation.Participants will be invited back to the lab 30 days (+/- 7 days) after the end of intervention to assess the longevity of any treatment effects.

ELIGIBILITY:
Inclusion Criteria:

1. children aged 11-16 years
2. With a confirmed diagnosis (wither clinical or genetic) of Neurofibromatosis Type 1
3. Informed consent/assent

Exclusion Criteria:

1. Child on active treatment for any NF1 related complications (such as chemotherapy for optic glioma)
2. Children with a known history of Epilepsy or on anti-epileptic medication
3. Children with poor verbal communication
4. Children with cardiac pacemakers, joint replacements or metal implants will be excluded.
5. Children with any previous operations to their head will be excluded.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
n-back test | Day 3 of intervention
  visuo-spatial and auditory n-back test to assess working memory

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Garg, MRCPsych, PhD, Principal Investigator — University of Manchester
Locations (1):
- University of Manchester, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
We plan to make the data available to other researchers upon request once the study has been completed.

REFERENCES:
- [Derived] Booth SJ, Garg S, Brown LJE, Green J, Pobric G, Taylor JR. Aberrant oscillatory activity in neurofibromatosis type 1: an EEG study of resting state and working memory. J Neurodev Disord. 2023 Aug 22;15(1):27. doi: 10.1186/s11689-023-09492-y. PMID 37608248